CLINICAL TRIAL: NCT05357677
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Crossover Study to Assess the Efficacy, Safety, and Tolerability of SR419 in Patients With Postherpetic Neuralgia (PHN)
Brief Title: To Evaluate the Efficacy and Safety of SR419 in Patients With Postherpetic Neuralgia (PHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai SIMR Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SR419-202
Record Dates: First submitted 2022-04-24; First posted 2022-05-03 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-03

CONDITIONS: Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SR419-Placebo sequence (Experimental): 30 mg of SR419 administered TID for 4 weeks followed by placebo administered TID for 4 weeks
  Interventions: Drug: SR419
- Placebo-SR419 sequence (Experimental): placebo administered TID for 4 weeks followed by 30 mg of SR419 administered TID for 4 weeks
  Interventions: Drug: SR419

INTERVENTIONS:
Drug: SR419 — SR419 capsule

SUMMARY:
This is a Phase II, international multicenter, double-blind, placebo-controlled, crossover study to assess the efficacy of SR419 in PHN subjects.

DETAILED DESCRIPTION:
The study will evaluate the efficacy and safety of SR419 in PHN patients. Each subject will participate in the study for up to approximately 14 weeks. This includes a screening period, drug treatment period, and post-treatment safety follow-up period. This is a crossover design study, in which subjects will be administered with SR419 and placebo according to their randomized sequence, that is, eligible subjects will be randomized in a 1:1 ratio to 1 of 2 double-blind treatment sequences: 30 mg of SR419 administered TID followed by placebo administered TID or placebo administered TID followed by 30 mg of SR419 administered TID.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female over 18 years old;
2. Having neuropathic pain of postherpetic neuralgia (PHN) that persists for >3 months after the herpes zoster rash is healed, with the pain area of a continuous area of affected rash.
3. DN4 score is ≥4 at Screening;
4. Average PI-NRS score of PHN-associated neuropathic pain over the last 24 hours at Screening is ≥4 and ≤9;
5. Female subjects must be non-pregnant and non-lactating;

Exclusion Criteria:

1. Other pains that cannot be clearly differentiated from PHN and may interfere with PHN assessment;
2. Circumstances that may affect pain assessment as determined by the investigator, such as skin disorders in the affected skin area that may affect sensation;
3. Active herpes zoster infection at screening;
4. Serious acute or chronic medical condition that, as assessed by the investigator, could increase the risks in subjects for participating in the trial or taking the study drug, or interfere with the study results;
5. Previous administration of other study drugs within 30 days or 5 half-lives before the study intervention used in this study (whichever is longer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Daily Average Pain Score (DAPS) | up to Day 64
  To assess the difference between the two treatment periods in the weekly average of Daily Average Pain Score (DAPS) at the last week. The pain intensity numerical rating scale (PI-NRS) consists of an 11-point numeric scale ranging from 0 (no pain) to 10 (worst imaginable pain). Participants described their pain during the past 24 hours by choosing the appropriate number between 0 and 10.

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGIC) | up to Day 64
  To assess the proportion of subjects who rate their pain as "much improved" or "very much improved" on the Patient Global Impression of Change (PGIC) at the end of each treatment period.
Daily Sleep Interference Score | up to Day 64
  To assess the within-subject difference between the two treatment periods in the weekly average of daily sleep interference scores at the last week. Pain-related sleep interference score was assessed on Daily Sleep Interference Scale (DSIS) which is an 11-point numerical rating scale ranging from 0 (did not interfere with sleep) to 10 (completely interfered [unable to sleep due to pain]). Participants were to describe how their pain had interfered with their sleep during the past 24 hours by choosing the appropriate number between 0 and 10.
Adverse events | up to Day 70
  To collect the adverse events during the study

OTHER OUTCOMES:
Plasma concentration of SR419 | on Day 15 and Day 36
  To measure the plasma concentration of SR419 after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Fa Bi Fan, MD, Principal Investigator — China-Japan Friendship Hospital; Yong Cui, MD, Principal Investigator — China-Japan Friendship Hospital
Locations (13):
- Australia (5):
  - PARC Clinical Research, Royal Adelaide Hospital, Adelaide
  - PARATUS Clinical Research Brisbane, Brisbane
  - PARATUS Clinical Research Canberra, Canberra
  - Genesis Research Services, Sydney
  - PARATUS Clinical Research Western Sydney, Sydney
- China (8):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing
  - Dermatology Hospital of Southern Medical University, Guangzhou
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Nanyang First People's Hospital, Nanyang
  - Huazhong University of Science and Technology Union Shenzhen Hospital, Shenzhen
  - The Second Hospital of Tianjin Medical University, Tianjin